CLINICAL TRIAL: NCT07118397
Title: Effect of Dry Needling Versus Kinesiology Taping in Patient With Plantar Fasciitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Anam Ashraf, physical therapist, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: anam.ashraf
Record Dates: First submitted 2025-07-31; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Plantar Fasciitis of Both Feet
Keywords: plantar fasciitis; Dry Needling, Kinesiology Taping; Heel Pain; Pain Management
MeSH Terms: conditions — Fasciitis, Plantar; Agnosia | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group/kinesiology taping (Experimental): The taping was applied for over 12 hours daily and was reapplied twice a week for a total of six weeks
  Interventions: Other: kinesiology taping
- group/dry needling (Experimental): Each dry needling session lasted for approximately 30 minutes. The total duration of the intervention was of 6 weeks with one session per week
  Interventions: Other: dry needling

INTERVENTIONS:
Other: dry needling — Dry needling involved the insertion of fine needles into identified myofascial trigger points within the plantar fascia and associated muscles. The technique aimed to release muscle tightness and alleviated pain by stimulating the trigger points. Needles were inserted perpendicularly to the skin at the identified trigger points, with the depth of insertion typically ranged from 35 to 70 mm, with 0.30mm diameter.
  Arms: group/dry needling
Other: kinesiology taping — Kinesiology Taping was applied using an I-shape technique. The taping began from the metatarsal head, extending through the plantar fascia and along the Achilles' tendon to the calf muscle. The application involved specific tension levels to support the plantar fascia and improve functional movement. The taping was applied with the foot in a slightly dorsiflexed position to ensure proper adherence and function.
  Arms: group/kinesiology taping

SUMMARY:
A single-blinded randomized controlled trial was conducted at hamza hospital Lahore ,Lahore poly clinic over 9 months. A total of 60 participants aged 20-45 years with clinically diagnosed plantar fasciitis and identifiable myofascial trigger points were recruited using a non-probability purposive sampling technique. They were randomly assigned to two groups (n=30 each): Group A received dry needling with conventional physiotherapy once per week, while Group B received kinesiology taping with conventional physiotherapy twice per week. Both interventions were administered for 6 weeks. Outcome measures included the Visual Analogue Scale (VAS) for pain, Foot and Ankle Outcome Score (FAOS) for functional assessment, and SF-12 Health Survey for quality of life. Assessments were conducted at baseline, week 3, and week 6.

DETAILED DESCRIPTION:
A single-blinded randomized controlled trial will be conducted at hamza hospital Lahore ,Lahore poly clinic. Total sixty patients aged 20-45 years with clinically diagnosed plantar fasciitis and identifiable myofascial trigger points. Group A received dry needling with conventional physiotherapy once per week, while Group B received kinesiology taping with conventional physiotherapy twice per week. Both interventions were administered for 6 weeks. Outcome measures included the Visual Analogue Scale (VAS) for pain, Foot and Ankle Outcome Score (FAOS) for functional assessment, and SF-12 Health Survey for quality of life. Assessments were conducted at baseline, week 3, and week 6.

ELIGIBILITY:
Inclusion Criteria:

* Participants age group included was 20 - 45 years (Al-Boloushi, 2019)
* Both genders were selected
* The presence of MTrPs on plantar and calf muscles was assured (Al-Boloushi, 2019)
* Patients with plantar fasciitis from less than 1 month Eftekharsadat, 2016)

Exclusion Criteria:

* Participants who have had an MTP injection 3 months before treatment (Yasar, 2021)
* Participants who have had fractures, Inflammatory joint or systemic disease, skin ulcers and neuropathy (Cotchett, 2014)
* Participants who have needle phobia (Al-Boloushi, 2019)
* Participants with history of prior foot or plantar surgery were excluded (Jianing, 2025)

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
plantar fasciitis | changes from pre -interventions to 6th week
  Plantar fasciitis is one of the most common causes of heel pain. It involves inflammation of a thick band of tissue that runs across the bottom of each foot and connects the heel bone to the toes, known as the plantar fascia
Pain Intensity | changes from pre interventions to 6th week
  Pain intensity will be measured using the Visual Analog Scale (VAS). The VAS is a continuous scale where participants indicate their pain level on a line ranging from 0 (no pain) to 10 (worst possible pain). The distance from the left end of the line to the participant's mark is measured in millimeters, providing a quantifiable score for pain intensity. A higher score reflects greater pain.
Functional Status | changes from pre -interventions to 6th week
  Functional status will be assessed using the Foot and Ankle Outcome Score (FAOS). The FAOS is a questionnaire designed to evaluate foot-related disability and pain, consisting of 13 items distributed across three domains: pain, disability, and activity limitation. Each item is rated from 0 (no problem) to 4 (severe problem). Scores for each domain are summed and averaged, with higher scores indicating worse functional status
Quality of Life(SF-12 ) | changes form pre-interventions to 6th week
  The SF-12 Health Survey will be used to assess quality of life. This tool evaluates physical and mental health outcomes, with scores reflecting overall well-being and daily functioning before and after treatment. The SF-12 provides a comprehensive measure of the impact of interventions on patients' quality of life. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamza Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Boloushi Z, Gomez-Trullen EM, Bellosta-Lopez P, Lopez-Royo MP, Fernandez D, Herrero P. Comparing two dry needling interventions for plantar heel pain: a protocol for a randomized controlled trial. J Orthop Surg Res. 2019 Jan 25;14(1):31. doi: 10.1186/s13018-019-1066-4. PMID 30683124